CLINICAL TRIAL: NCT05448872
Title: Real World Experience in HFrEF Patients Treated With sAc/vaL in ITaly
Brief Title: Real World Experience in Heart Failure With Reduced Ejection Fraction (HFrEF) Patients Treated With sAc/vaL.
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLCZ696BIT08
Record Dates: First submitted 2022-07-01; First posted 2022-07-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Heart Failure
Keywords: Drug utilization,; Heart failure,; Real-world,; Sacubitril/Valsartan
MeSH Terms: conditions — Heart Failure | interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Sacubitril/Valsartan: Heart Failure (HF) patients treated with Sac/Val
  Interventions: Drug: Sacubitril/Valsartan

INTERVENTIONS:
Drug: Sacubitril/Valsartan — HF patients treated with Sac/Val

SUMMARY:
The study is a cohort observational, retrospective, non-interventional study.

DETAILED DESCRIPTION:
Study period:

Index date: The index date were defined as the first date of the first prescription of Sacubitril/Valsartan during inclusion period and this were used to establish the beginning of the follow-up period.

Characterization period: 6 months period before the index date were used to characterize patients.

Follow-up period: Any patients has at least 1 year of follow-up. Follow-up period went from index date to June 2020.

ELIGIBILITY:
Inclusion Criteria:

Consecutive ambulatory patients with a diagnosis of HF that attended the Outpatient Clinics for HF management and who have been prescribed Sacubitril/Valsartan from 01 October 2016 to 30 June 2019 (inclusion period) were included in the study. To allow for at least 1-year follow-up period for any patients, the observation period ended by 30 June 2020.

In detail, all patients attending by outpatient clinics for the diagnosis and treatment of HF in the Italian Centers involved, with:

* age ≥18 years old AND
* at least one prescription of Sacubitril/Valsartan from 01 October 2016 to 30 June 2019 were included in the study.

Exclusion Criteria:

* Missing age or sex information.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart Failure with reduced Ejection Fraction (HfrEF) patients treated with Sacubitril/Valsartan.
Sampling Method: Non-Probability Sample
Enrollment: 924 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Age | Baseline
  To describe the demographics
Gender | Baseline
  To describe the demographics
Number of patients with Ischemic heart disease | Baseline
  To evaluate clinical characteristics at baseline.
Number of patients with PCI/CABG: Percutaneous coronary intervention/coronary artery bypass grafting | Baseline
  To evaluate clinical characteristics at baseline.
Number of patients with moderate or severe mitral or aortic valvulopathy | Baseline
  To evaluate clinical characteristics at baseline.
Number of patients with Implanted prosthetic valve | Baseline
  To evaluate clinical characteristics at baseline.
Number of patients with ICD/CRT, Implantable Cardioverter Defibrillator/ Cardiac Resynchronization Therapy | Baseline
  To evaluate clinical characteristics at baseline.
Number of patients with Atrial fibrillation | Baseline
  To evaluate clinical characteristics at baseline.
Number of patients with prior hospitalization for HF | Baseline
  To evaluate clinical characteristics at baseline.
Number of patients with previous stroke | Baseline
  To evaluate clinical characteristics at baseline.
Number of patients with diabetes mellitus | Baseline
  To evaluate clinical characteristics at baseline.
Number of patients with Hypertension | Baseline
  To evaluate clinical characteristics at baseline.
Number of patients with Chronic kidney disease (CKD) | Baseline
  To evaluate clinical characteristics at baseline.
Duration of HF disease | Baseline
  To evaluate clinical characteristics at baseline.
Number of patients with pharmacological treatments for HF | throughout the study, approximately 3 years
  To evaluate the pharmacological treatments for HF during characterization and follow-up.

SECONDARY OUTCOMES:
Number of patients with initial and final doses | throughout the study, approximately 3 years
  To evaluate the Sacubitril/Valsartan dosing pattern during follow-up
Number of patients with Non-maximum dose | throughout the study, approximately 3 years
  To evaluate the Sacubitril/Valsartan dosing pattern during follow-up
Time to maximal dose prescribed | throughout the study, approximately 3 years
  To evaluate the Sacubitril/Valsartan dosing pattern during follow-up
Number of patients with hospitalization HF-related | throughout the study, approximately 3 years
  To evaluate frequency of cardiovascular (CV) and non-CV death.
Number of patients with hospitalization related to other cardiovascular events | throughout the study, approximately 3 years
  To evaluate frequency of cardiovascular (CV) and non-CV death.
Number of patients with hospitalization related to non-CV cause | throughout the study, approximately 3 years
  To evaluate frequency of cardiovascular (CV) and non-CV death.
Number of patients with Percutaneous Coronary Intervention (PCI)/coronary artery bypass grafting (CABG) | throughout the study, approximately 3 years
  To evaluate frequency of cardiovascular (CV) and non-CV death.
Number of patients with Valvular intervention | throughout the study, approximately 3 years
  To evaluate frequency of cardiovascular (CV) and non-CV death.
Number of patients with Device implantation (ICD/CRT) | throughout the study, approximately 3 years
  To evaluate frequency of cardiovascular (CV) and non-CV death.
Number of patients with ER visits HF-related | throughout the study, approximately 3 years
  To evaluate frequency of cardiovascular (CV) and non-CV death.
Number of deaths | throughout the study, approximately 3 years
  To evaluate frequency of cardiovascular (CV) and non-CV death.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Trieste, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for CLCZ696BIT08 from the Novartis Clinical Trials Website — http://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17954